CLINICAL TRIAL: NCT02817516
Title: A Randomized, Double-Blind (Sponsor-Open), Placebo-Controlled, Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Escalating Multiple Doses of TAK-828 in Healthy Subjects
Brief Title: A Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics Study of TAK-828 Escalating Multiple-Doses in Healthy Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: TAK-828-1002; U1111-1177-8105 (Registry Identifier: WHO)
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Results first posted 2019-07-17 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-04

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- Part 1: TAK-828 15 milligram (mg) (Experimental): TAK-828 15 mg, solution (0.2 milligram per milliliter [mg/mL] or 5 mg/mL), orally, twice daily on Days 1-13, and once on the morning of Day 14 in healthy non-Japanese participants.
  Interventions: Drug: TAK-828
- Part 1: TAK-828 45 mg (Experimental): TAK-828 45 mg, solution (0.2 mg/mL or 5 mg/mL), orally, twice daily on Days 1-13, and once on the morning of Day 14 in healthy non-Japanese participants.
  Interventions: Drug: TAK-828
- Part 1: TAK-828 75 mg (Experimental): TAK-828 75 mg, solution (0.2 mg/mL or 5 mg/mL), orally, twice daily on Days 1-13, and once on the morning of Day 14 in healthy non-Japanese participants.
  Interventions: Drug: TAK-828
- Part 1: TAK-828 100 mg (Experimental): TAK-828 100 mg, solution (0.2 mg/mL or 5 mg/mL), orally, twice daily on Days 1-13, and once on the morning of Day 14 in healthy non-Japanese participants.
  Interventions: Drug: TAK-828
- Part 2: TAK-828 45 mg (Experimental): TAK-828 45 mg, solution (0.2 mg/mL or 5 mg/mL), orally, twice daily on Days 1-13, and once on the morning of Day 14 in healthy Japanese participants.
  Interventions: Drug: TAK-828
- Part 2: TAK-828 100 mg (Experimental): TAK-828 100 mg, solution (0.2 mg/mL or 5 mg/mL), orally, twice daily on Days 1-13, and once on the morning of Day 14 in healthy Japanese participants.
  Interventions: Drug: TAK-828
- Part 1: Placebo (Placebo Comparator): TAK-828 placebo-matching solution, orally, twice daily on Days 1-13, and once on the morning of Day 14 in healthy non-Japanese participants.
  Interventions: Drug: Placebo
- Part 2: Placebo (Placebo Comparator): TAK-828 placebo-matching solution, orally, twice daily on Days 1-14 in healthy Japanese participants.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAK-828 — TAK-828 solution.
  Arms: Part 1: TAK-828 100 mg; Part 1: TAK-828 15 milligram (mg); Part 1: TAK-828 45 mg; Part 1: TAK-828 75 mg; Part 2: TAK-828 100 mg; Part 2: TAK-828 45 mg
Drug: Placebo — TAK-828 placebo-matching solution.
  Arms: Part 1: Placebo; Part 2: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of multiple oral doses of TAK-828 in healthy participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-828. TAK-828 is being tested to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics in healthy non-Japanese and Japanese participants in Parts 1 and 2, respectively.

The study will enroll approximately 56 participants. Participants will be randomly assigned (by chance, like flipping a coin) to receive either TAK-828 or matching placebo. This assignment will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need).

Proposed doses:

* Part 1: TAK-828 15 mg, 45 mg, 75 mg, 100 mg, and placebo twice daily
* Part 2: TAK-828 45 mg, and 100 mg, and placebo twice daily

All participants will be asked to take the solution at the same time each day throughout the study.

This multi-center trial will be conducted in the United States.

ELIGIBILITY:
Inclusion:

For Parts 1 and 2, participant eligibility is determined according to the following criteria prior to entry into the study:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative, signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures including requesting that a participant fast for any laboratory evaluations.
3. The participant is a healthy male, or a healthy female not of child-bearing potential. Females not of childbearing potential are defined as those who have been surgically sterilized (hysterectomy, bilateral oophorectomy or tubal ligation) or who are postmenopausal (example, defined as at least 1 year since last regular menses, with a follicle-stimulating hormone [FSH] level of greater than (>) 40 international units per liter [IU/L] or at least 5 years since last regular menses confirmed before any study drug is administered).
4. For Part 1: the participant is a non-Japanese adult, aged 18 to 55 years (inclusive) at the time of informed consent and first dose of study drug.
5. For Part 1: the participant weighs at least 50 kilogram (kg) and has a body mass index (BMI) of 18 to 30 kilogram per square meter (kg/m^2) (inclusive) at Screening.
6. For Part 2: the participant is of Japanese descent (born to Japanese parents and grandparents), aged 20 to 55 years (inclusive) at the time of informed consent and first dose of study drug.
7. For Part 2: the participant weighs at least 45 kg and has a BMI of 18.5 to 25 kg/m^2 (inclusive) at Screening.

Exclusion Criteria

For Parts 1 and 2, any participant who meets any of the following criteria will not qualify for entry into the study:

1. The participant received any investigational compound within 30 days or 5 half-lives (whichever is longer) before the first dose of study drug.
2. The participant used prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) before Check-in (Day -1). Herbal supplements and hormone replacement therapy (HRT) must be discontinued 28 days prior to Check-in (Day -1). As an exception, acetaminophen may be used at doses of less than or equal to (<=) 1 gram/day. Limited use of nonprescription medications that are not believed to affect participant safety or the overall results of the study may be permitted on a case-by-case basis following approval by the sponsor.
3. The participant is an immediate family member or study-site employee or is in a dependent relationship with a study-site employee who is involved in the conduct of this study (example, spouse, parent, child, sibling) or may consent under duress.
4. The participant has a history or presence of any disease or condition (or there is any finding upon review of the participant's medical history, physical examination, or clinical laboratory tests giving reasonable suspicion of a disease) that could interfere with study participation or safety, contraindicate taking TAK-828 or a similar drug in the same class, or potentially confound the study results (example, history or presence of clinically significant neurologic, cardiovascular, pulmonary, hepatic, hematologic, renal, immunologic, metabolic, musculoskeletal, gastrointestinal, endocrine, or psychiatric disease). It is the responsibility of the investigator to assess the clinical significance; however, consultation with the Takeda medical monitor may be warranted.
5. The participant has a known hypersensitivity to any component of the formulation of TAK-828.
6. The participant has an active infection at Screening.
7. The participant has a positive urine drug result for drugs of abuse (defined as any illicit drug use) at Screening or Check-in (Day -1).
8. The participant has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year, or the participant drinks 7 or more drinks/week for females or 14 or more drinks/week for males (1 drink=5 ounces [150 milliliter {mL}] of wine, 12 ounces [360 mL] of beer, or 1.5 ounces [45 mL] of hard liquor) within 6 months before the Screening visit or is unwilling to abstain from alcohol and drugs throughout the study.
9. The participant is taking or took any excluded medication, supplements, or food products during the time periods listed in the Prohibited Medications, Foods, and Products table
10. If male, the participant intends to donate sperm during the course of this study or for 14 weeks after the last dose of study drug.
11. The participant has any condition possibly affecting drug absorption (example, gastrectomy).
12. The participant has a history of cancer, except basal cell carcinoma that has been in remission for at least 5 years before Screening.
13. The participant has a positive test result for hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibody at Screening or has a known history of human immunodeficiency virus (HIV) infection.
14. The participant used nicotine-containing products (including, but not limited to, cigarettes, pipes, cigars, chewing tobacco, nicotine patch, or nicotine gum) within 28 days prior to Check-in (Day -1) or cotinine test is positive at Screening or Check-in (Day -1).
15. The participant has poor peripheral venous access.
16. The participant donated or lost 450 mL or more of his or her blood volume (including plasmapheresis) or had a transfusion of any blood product within 30 days prior to Day 1.
17. The participant has a Screening or Check-in (Day -1) abnormal (clinically significant) ECG. Entry of any participant with an abnormal (not clinically significant) ECG must be approved, and documented by signature of the principal investigator or medically qualified subinvestigator.
18. The participant has abnormal Screening or Day -1 laboratory values that suggest a clinically significant underlying disease or the participant has the following laboratory abnormalities: alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 3 times the upper limit of normal (ULN).
19. The participant has a creatine kinase isoenzyme MB (CK-MB) or cardiac troponin above the ULN at Screening or Day -1.
20. If female, the participant is of childbearing potential (example, premenopausal, not sterilized).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2016-08-22 (Actual); Study Completion 2016-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/Approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 30 June 2016 to 22 August 2016.
Pre-assignment Details: Non-Japanese healthy participants were enrolled in Part 1 to receive TAK-828 as multiple rising dose of: 15 milligram (mg) in Cohort 1, 45 mg in Cohort 2, and 75 mg in Cohort 3. Study was terminated before the start of 100 mg in Part 1 Cohort 4, and 45 mg and 100 mg in Japanese participants in Part 2 due to findings from 13-week toxicology study.
Groups:
- Part 1 Cohorts 1 to 3: Placebo: TAK-828 placebo-matching solution, orally, twice daily on Days 1 to 13, and once in the morning of Day 14 in healthy non-Japanese participants.
- Part 1 Cohort 1: TAK-828 15 mg: TAK-828 15 mg, solution (0.2 milligram per milliliter [mg/mL] or 5 mg/mL), orally, twice daily on Days 1 to 13, and once in the morning of Day 14 in healthy non-Japanese participants.
- Part 1 Cohort 2: TAK-828 45 mg: TAK-828 45 mg, solution (0.2 mg/mL or 5 mg/mL), orally, twice daily on Days 1 to 13, and once in the morning of Day 14 in healthy non-Japanese participants.
- Part 1 Cohort 3: TAK-828 75 mg: TAK-828 75 mg, solution (0.2 mg/mL or 5 mg/mL), orally, twice daily on Days 1 to 13, and once in the morning of Day 14 in healthy non-Japanese participants.
Period: Overall Study
Arm/Group | Part 1 Cohorts 1 to 3: Placebo | Part 1 Cohort 1: TAK-828 15 mg | Part 1 Cohort 2: TAK-828 45 mg | Part 1 Cohort 3: TAK-828 75 mg
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 5 | 6
Not Completed | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety set included all participants who received at least 1 dose of study drug.
Groups:
- Part 1 Cohort 1: TAK-828 15 mg: TAK-828 15 mg, solution (0.2 mg/mL or 5 mg/mL), orally, twice daily on Days 1 to 13, and once in the morning of Day 14 in healthy non-Japanese participants.
- Total: Total of all reporting groups
Arm/Group | Part 1 Cohorts 1 to 3: Placebo | Part 1 Cohort 1: TAK-828 15 mg | Part 1 Cohort 2: TAK-828 45 mg | Part 1 Cohort 3: TAK-828 75 mg | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (7.78) | 40.3 (8.45) | 26.5 (3.73) | 37.0 (14.63) | 34.8 (10.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 0 | 2
  Male | 5 | 5 | 6 | 6 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3 | 4 | 10
  Not Hispanic or Latino | 6 | 3 | 3 | 2 | 14
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 1 | 0 | 4
  White | 2 | 5 | 3 | 6 | 16
  More than one race | 0 | 0 | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 6 | 6 | 24
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 172.3 (11.72) | 171.8 (9.15) | 175.3 (2.42) | 168.5 (3.94) | 172.0 (7.67)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 77.75 (15.209) | 72.23 (6.696) | 77.45 (9.702) | 73.45 (11.232) | 75.22 (10.679)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 25.97 (2.645) | 24.48 (1.525) | 25.17 (2.743) | 25.87 (3.974) | 25.37 (2.733)
Smoking Classification [Count of Participants; unit: Participants]
  Never smoked | 5 | 5 | 5 | 4 | 19
  Ex-smoker | 1 | 1 | 1 | 2 | 5
Alcohol Classification [Count of Participants; unit: Participants]
  Never drunk | 5 | 2 | 3 | 3 | 13
  Current drinker | 1 | 2 | 2 | 2 | 7
  Ex-drinker | 0 | 2 | 1 | 1 | 4
Caffeine/Xanthine Consumption [Count of Participants; unit: Participants]
  Had caffeine/xanthine consumption | 1 | 2 | 2 | 4 | 9
  Had no caffeine/xanthine consumption | 5 | 4 | 4 | 2 | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experience at Least One Treatment Emergent Adverse Event (TEAE)
Time Frame: Baseline up to 10 days after last dose of study drug (Day 24)
Population: The safety set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 Cohorts 1 to 3: Placebo | Part 1 Cohort 1: TAK-828 15 mg | Part 1 Cohort 2: TAK-828 45 mg | Part 1 Cohort 3: TAK-828 75 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
percentage of participants | 16.7 | 33.3 | 50.0 | 16.7

2. Primary Outcome: Percentage of Participants Who Discontinued the Treatment Due to an Adverse Event (AE)
Time Frame: Baseline up to 10 days after last dose of study drug (Day 24)
Population: The safety set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 Cohorts 1 to 3: Placebo | Part 1 Cohort 1: TAK-828 15 mg | Part 1 Cohort 2: TAK-828 45 mg | Part 1 Cohort 3: TAK-828 75 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
percentage of participants | 0 | 0 | 0 | 0

3. Primary Outcome: Percentage of Participants Who Meet the Markedly Abnormal Criteria for Safety Laboratory Tests at Least Once Post-dose
Time Frame: Baseline up to 10 days after last dose of study drug (Day 24)
Population: The safety set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 Cohorts 1 to 3: Placebo | Part 1 Cohort 1: TAK-828 15 mg | Part 1 Cohort 2: TAK-828 45 mg | Part 1 Cohort 3: TAK-828 75 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
percentage of participants | 0 | 0 | 0 | 0

4. Primary Outcome: Percentage of Participants Who Meet the Markedly Abnormal Criteria for Vital Sign Measurements at Least Once Post-dose
Time Frame: Baseline up to 10 days after last dose of study drug (Day 24)
Population: The safety set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 Cohorts 1 to 3: Placebo | Part 1 Cohort 1: TAK-828 15 mg | Part 1 Cohort 2: TAK-828 45 mg | Part 1 Cohort 3: TAK-828 75 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
percentage of participants
  Systolic blood pressure (BP) supine <85 mmHg | 0 | 16.7 | 0 | 0
  Systolic BP standing<85millimeter of mercury(mmHg) | 16.7 | 0 | 0 | 0
  Diastolic BP supine less than (<) 50 mm Hg | 0 | 16.7 | 0 | 0
  Diastolic BP standing <50 mm Hg | 0 | 0 | 16.7 | 0
  Pulse rate supine <50 beats per minute (bpm) | 16.7 | 0 | 0 | 0
  Pulse rate 5 minutes supine <50 bpm | 16.7 | 33.3 | 50.0 | 50.0
  Pulse rate 1 minute standing <50 bpm | 16.7 | 0 | 0 | 0
  Pulse rate 3 minute standing <50 bpm | 16.7 | 0 | 0 | 0
  Pulse rate 3 minute standing greater than 120 bpm | 0 | 16.7 | 0 | 0
  Temperature <35.6 Celsius | 0 | 0 | 33.3 | 33.3

5. Primary Outcome: Percentage of Participants Who Meet the Markedly Abnormal Criteria for Safety 12-lead Electrocardiogram (ECG) at Least Once Post-dose
Time Frame: Baseline up to 10 days after last dose of study drug (Day 24)
Population: The safety set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 Cohorts 1 to 3: Placebo | Part 1 Cohort 1: TAK-828 15 mg | Part 1 Cohort 2: TAK-828 45 mg | Part 1 Cohort 3: TAK-828 75 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
percentage of participants
  Heart Rate <50 bpm | 16.7 | 33.3 | 33.3 | 50.0
  QT Interval greater than or equalto 460millisecond | 16.7 | 0 | 16.7 | 0

6. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for Free Base of TAK-828 (TAK-828F)
Time Frame: Days 1 and 7 pre-dose and at multiple time points (up to 24 hours) post-dose and Day 14 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: Pharmacokinetic (PK) set included all participants who received at least 1 dose of study drug, had at least 1 measurable plasma/urine concentration of TAK-828F. PK set where data at specified time points was available. PK data was not collected for Day 7 and 14 Part 1 Cohort 3, as participants received last dose on Day 6 due to study termination.
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part 1 Cohort 1: TAK-828 15 mg | Part 1 Cohort 2: TAK-828 45 mg | Part 1 Cohort 3: TAK-828 75 mg
Number analyzed (Participants) | 6 | 6 | 6
nanogram per milliliter (ng/mL)
  Day 1: number analyzed (Participants) | 6 | 5 | 6
  Day 1 | 1170 (302) | 3750 (562) | 9680 (1580)
  Day 7: number analyzed (Participants) | 6 | 5 | 0
  Day 7 | 1480 (230) | 4610 (619) |
  Day 14: number analyzed (Participants) | 6 | 5 | 0
  Day 14 | 1310 (345) | 4600 (524) |

7. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-828F
Time Frame: as for outcome 6
Population: PK set included all participants who received at least 1 dose of study drug, had at least 1 measurable plasma/urine concentration of TAK-828F. PK set where data at specified time points was available. PK data was not collected for Day 7 and 14 Part 1 Cohort 3, as participants received last dose on Day 6 due to study termination.
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1 Cohort 1: TAK-828 15 mg | Part 1 Cohort 2: TAK-828 45 mg | Part 1 Cohort 3: TAK-828 75 mg
Number analyzed (Participants) | 6 | 6 | 6
hours
  Day 1: number analyzed (Participants) | 6 | 5 | 6
  Day 1 | 1.0 [0.5 to 2.0] | 1.0 [0.5 to 1.0] | 1.0 [0.5 to 2.05]
  Day 7: number analyzed (Participants) | 6 | 5 | 0
  Day 7 | 1.0 [0.5 to 2.05] | 0.5 [0.5 to 1.0] |
  Day 14: number analyzed (Participants) | 6 | 5 | 0
  Day 14 | 1.0 [0.5 to 1.0] | 0.5 [0.5 to 1.0] |

8. Secondary Outcome: AUCtau: Area Under the Plasma Concentration-time Curve From Time 0 to Time Tau Over the Dosing Interval for TAK-828F
Time Frame: Cohorts 1 and 2: Days 1 and 7 pre-dose and at multiple time points (up to 24 hours) post-dose and Day 14 pre-dose and at multiple time points (up to 72 hours) post-dose; Cohort 3: Day 1 pre-dose and at multiple time points (up to 24 hours) post-dose
Population: as for outcome 7
Measure: Geometric Mean (Standard Deviation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Part 1 Cohort 1: TAK-828 15 mg | Part 1 Cohort 2: TAK-828 45 mg | Part 1 Cohort 3: TAK-828 75 mg
Number analyzed (Participants) | 6 | 6 | 6
hour*nanogram per milliliter (h*ng/mL)
  Day 1: number analyzed (Participants) | 6 | 5 | 6
  Day 1 | 5090 (1300) | 15400 (1360) | 40000 (5870)
  Day 7: number analyzed (Participants) | 6 | 5 | 0
  Day 7 | 6730 (1320) | 17900 (3060) |
  Day 14: number analyzed (Participants) | 6 | 5 | 0
  Day 14 | 6890 (1540) | 20600 (3860) |

ADVERSE EVENTS:
Time Frame: TEAEs are adverse events that started after the first dose of double-blind study drug and no more than 10 days (Day 24) after the last dose of double-blind study drug
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Part 1 Cohorts 1 to 3: Placebo | Part 1 Cohort 1: TAK-828 15 mg | Part 1 Cohort 2: TAK-828 45 mg | Part 1 Cohort 3: TAK-828 75 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/6 | 2/6 | 3/6 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Cohorts 1 to 3: Placebo (N=6) | Part 1 Cohort 1: TAK-828 15 mg (N=6) | Part 1 Cohort 2: TAK-828 45 mg (N=6) | Part 1 Cohort 3: TAK-828 75 mg (N=6)
Dry eye (Eye disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.